CLINICAL TRIAL: NCT00967148
Title: The Use of Extended Perioperative Low Molecular Weight Heparin to Improve Cancer Specific Survival Following Surgical Resection of Colon Cancer: A Pilot Randomized Controlled Trial
Brief Title: Thromboprophylaxis for Patients Undergoing Surgical Resection for Colon Cancer
Acronym: PERI-OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009121-01H
Record Dates: First submitted 2009-07-08; First posted 2009-08-27 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism; Cancer
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Neoplasms | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tinzaparin (Experimental): The treatment arm will receive a subcutaneous injection of tinzaparin (4500U) daily beginning within two days of the decision to operate (within 6 weeks of surgical resection) weeks and continued for 4 weeks following resection.
  Interventions: Drug: Tinzaparin
- Standard of care (Active Comparator): The control arm will receive a subcutaneous injection of 4,500 U of tinzaparin daily beginning with the first postoperative dose and continued for the duration of hospitalization.
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — The treatment arm will receive a subcutaneous injection of tinzaparin (4500U) daily beginning within two days of the decision to operate (within 6 weeks of surgical resection) weeks and continued for 4 weeks following resection.
  Other Names: Innohep

SUMMARY:
The blood thinner "tinzaparin" might increase survival in patients with colon cancer undergoing surgical resection. The investigators want to assess if a trial allocating patients to prolonged treatment with tinzaparin versus standard of care is feasible.

DETAILED DESCRIPTION:
Cancer patients are at high risk of postoperative thrombosis and this risk remains elevated beyond the period of hospitalization. Thromboprophylaxis effectively reduces the risk of post operative VTE in cancer patients. Extended thromboprophylaxis beyond hospitalization (up to 30 days) with LMWH has been shown to further reduce the risk of postoperative VTE. Concurrently, there is a growing body of evidence to suggest that LMWH may have anti-cancer effects due to anti-metastatic properties and may improve survival in cancer patients, even in the absence of a documented VTE. Retrospective studies have shown that perioperative thromboprophylaxis (i.e., starting thromboprophylaxis before the surgery) seems to increase survival in cancer patients undergoing abdominal or pelvic cancer surgery with curative intent. The investigators propose to perform an open-label RCT to determine if thromboprophylaxis using tinzaparin 4,500 IU daily, starting from the time of decision to operate through the peri-operative period and extending for 4 weeks postoperatively, is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older with a pathologically confirmed localized invasive colorectal cancer and no evidence of metastatic disease who are scheduled to undergo surgical resection will be eligible.
* All study patients must be enrolled at least two weeks prior to scheduled surgery and provide written informed consent.
* All the following criteria must be met to be eligible:

  1. Pathological confirmation of an invasive adenocarcinoma of the colon;
  2. No evidence of metastatic disease by Computed Tomography (CT) scan of the abdomen and pelvis or chest X-ray (CXR). A Magnetic Resonance Imaging (MRI) of the abdomen and pelvis will be used if the patient has a documented contrast allergy or to verify a questionable finding on the CT scan. Any abnormal findings on CXR will be investigated with a CT scan of the chest. Imaging must be performed within 2 months of randomization;
  3. a scheduled surgical operation for resection of the colon cancer; and
  4. ECOG performance status 0 or 1.

Exclusion Criteria:

* Subjects cannot be included in this study if any of the following criteria apply:

  1. rectal adenocarcinoma (defined as tumor below the peritoneal reflection or within 12 cm of the anal verge by rigid sigmoidoscopy);
  2. prior VTE including deep vein thrombosis (DVT) or pulmonary embolism (PE);
  3. requirement for full dose perioperative anticoagulation;
  4. requirement for anti-platelet or anti-inflammatory therapy that cannot be discontinued;
  5. contraindication to heparin therapy **;
  6. geographic inaccessibility (less likely to comply with required follow-up visits and care);
  7. participating in another interventional trial that may result in co-intervention or contamination (to be determined by PI);
  8. < 18 years of age;
  9. history of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within 5 years of the colorectal cancer diagnosis;
  10. treatment, including radiation therapy, chemotherapy or targeted therapy, administered for the currently diagnosed colon cancer prior to randomization;
  11. pregnant or lactating; and
  12. unable/unwilling to providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 3 months

SECONDARY OUTCOMES:
Refusal rate | 3 months
Rate of non-compliance and lost to follow-up | 6 months
Expression of sialylated fucosylated glycans (including CA19-9, sialyl Lewis X and CD24) in primary tumor specimens by immunohistochemistry (IHC). | postoperative day 0, 1, 4, 7±1, and 28±4
Expression of TF. VEGF and microvessel density in primary tumor specimens by IHC. | postoperative day 0, 1, 4, 7±1, and 28±4
Serum soluble TF and TFPI levels pre and postoperatively (postoperative day 0, 1, 4, 7±1, and 28±4) measured by enzyme linked immunosorbent assay (ELISA). | postoperative day 0, 1, 4, 7±1, and 28±4
Platelet count and serum soluble P-selectin levels pre and postoperatively (postoperative day 0, 1, 4, 7±1, and 28±4) measured by hemocytometer and ELISA. | postoperative day 0, 1, 4, 7±1, and 28±4
Serum VEGF levels pre and postoperatively (postoperative day 0, 1, 4, 7±1, and 28±4) measured by ELISA | postoperative day 0, 1, 4, 7±1, and 28±4
Quantification and characterization of VPC pre and postoperatively (postoperative day 0, 1, 4, 7±1, and 28±4) measured by VPC cell culture assay and flow cytometry. | postoperative day 0, 1, 4, 7±1, and 28±4

CONTACTS AND LOCATIONS:
Overall Officials: Marc Carrier, MD MSc, Principal Investigator — Ottawa Hospital Research Institute; Rebecca Auer, MD MSc, Principal Investigator — Ottawa Hospital Research Institute; Tim Asmis, MD, Study Chair — Ottawa Hospital
Locations (1):
- Ottawa Health Research Institute, Ottawa, Ontario, Canada